CLINICAL TRIAL: NCT02806570
Title: Early Feasibility Study of the AccuCinch® Ventricular Restoration System
Brief Title: The CorCinch - Functional Mitral Valve Regurgitation (FMR) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ancora Heart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 4433
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Mitral Valve Insufficiency; Cardiomyopathies
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency; Cardiomyopathies | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AccuCinch® Ventricular Restoration System (Experimental)
  Interventions: Device: Mitral valve repair

INTERVENTIONS:
Device: Mitral valve repair

SUMMARY:
This is a multi-center, non-randomized, prospective Early Feasibility Study to evaluate the AccuCinch® Ventricular Restoration System in patients with symptomatic heart failure and concomitant functional mitral regurgitation that have stable symptoms on guideline-directed medical therapy

DETAILED DESCRIPTION:
Device name changed from AccuCinch® Ventricular Repair System to AccuCinch® Ventricular Restoration System, FDA Approval Date 08Aug2020

ELIGIBILITY:
Inclusion Criteria:

* Study patient is at least 18-years old
* Severity of FMR: ≥ Moderate (i.e., 2+, according to Stone et al Clinical Trial Design Principles and Endpoint Definitions for Transcatheter Mitral Valve Repair and Replacement: Part 1: Clinical Trial Design Principles. A Consensus Document from the Mitral Valve Academic Research Consortium11; and 2003 ASE Guidelines for grading mitral regurgitation10)
* Ejection Fraction: ≥20 to ≤60%
* Symptom Status: NYHA II-IV (i.e., ambulatory)
* Treatment and compliance with optimal guideline directed medical therapy for heart failure for at least 1 month
* Surgical risk: Subject is eligible for cardiac surgery (specific risk score or comorbidities should demonstrate high risk features, as determined by the Heart Team)
* Completion of all qualifying diagnostic and functional tests and agrees to comply with study follow-up schedule

Exclusion Criteria:

* Patients with significant organic mitral valve pathology (e.g. myxomatous degeneration, mitral valve prolapse or flail leaflets)
* Myocardial infarction or any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
* Prior surgical, transcatheter, or percutaneous mitral valve intervention
* Untreated clinically significant coronary artery disease (CAD) requiring revascularization
* Hemodynamic instability: Hypotension (systolic pressure <90 mmHg) or requirement for inotropic support or mechanical hemodynamic support
* Any planned cardiac surgery or interventions within the next 6 months (including right heart procedures)
* NYHA class IV (i.e., non-ambulatory) or American College of Cardiology (ACC)/American Heart Association (AHA) Stage D heart failure
* Fixed pulmonary artery systolic pressure >70 mmHg
* Severe tricuspid regurgitation (per ASE guidelines and graded by the Echo Core Lab)
* Modified Rankin Scale ≥ 4 disability
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
* Anatomical pathology/constraints preventing appropriate access/implant of the AccuCinch® Ventricular Restoration System (e.g., femoral arteries will not support a 20F system)
* Renal insufficiency (i.e., eGFR of <30ml/min/1.73m2; Stage 4 or 5 CKD)
* Moderate or severe aortic valve stenosis or regurgitation or aortic valve prosthesis
* Fluoroscopic or echocardiographic evidence of severe aortic arch calcification, mobile aortic atheroma, intracardiac mass, thrombus or vegetation
* Active bacterial endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
30-Day Safety | 30-day
  Assess 30-day safety defined as device-related or procedure-related major adverse events (MAEs).
  MAE is a composite of death; myocardial infarction; emergent conversion to surgery; stroke; major cardiac structure complication; major vascular complication; and heart failure-related hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zapien, MS, CCRA, Study Director — Ancora Heart, Inc. (formerly Guided Delivery Systems Inc.); Dean Kereiakes, MD, Principal Investigator — The Christ Hospital; Satya Shreenivas, MD, Principal Investigator — The Christ Hospital
Locations (16):
- United States (16):
  - Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Minneapolis Heart Foundation Institute, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute / Nebraska Heart Hospital, Lincoln, Nebraska
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Baylor College of Medicine St. Luke's Medical Center, Houston, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - University of Washington Medicine, Seattle, Washington